CLINICAL TRIAL: NCT03070184
Title: Racial Differences in the Natriuretic Peptide Response to Exercise and Beta-blockers
Brief Title: Race, Natriuretic Peptides and Physiological Perturbations
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Pankaj Arora, MD, Associate Professor, University of Alabama at Birmingham
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: IRB-170214001; K23HL146887 (NIH)
Record Dates: First submitted 2017-02-28; First posted 2017-03-03 (Actual); Results first posted 2025-02-27 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Healthy; Pre Hypertension
Keywords: Racial differences
MeSH Terms: conditions — Prehypertension | interventions — Metoprolol

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Black Participants (Experimental): Healthy lean (BMI 18-25 kg/m2) African-American participants will be enrolled and each will undergo a physical exam and screening tests to determine participants' eligibility. Participants will perform exercise capacity VO2 max determination test, followed by 3 days of standardized meals and exercise challenge test. After exercise challenge test, all the participants will receive metoprolol succinate starting at 50mg/day, titrated bi-weekly up to 200 mg/day.
  Interventions: Other: Exercise capacity VO2 max determination; Dietary Supplement: Standardized meals; Other: Exercise challenge; Drug: Metoprolol Succinate ER
- White Participants (Active Comparator): Healthy lean (BMI 18-25 kg/m2) white participants will be enrolled and each will undergo a physical exam and screening tests to determine participants' eligibility. Participants will perform exercise capacity VO2 max determination test, followed by 3 days of standardized meals and exercise challenge test. After exercise challenge test, all the participants will receive metoprolol succinate starting at 50mg/day, titrated bi-weekly up to 200 mg/day.
  Interventions: Other: Exercise capacity VO2 max determination; Dietary Supplement: Standardized meals; Other: Exercise challenge; Drug: Metoprolol Succinate ER

INTERVENTIONS:
Other: Exercise capacity VO2 max determination — Each participant's maximal oxygen capacity will be determined using a modified Bruce treadmill protocol.
Dietary Supplement: Standardized meals — Participants will consume the standardized study diet for 3 days provided by the clinical research unit's metabolic kitchen (at UAB).
Other: Exercise challenge — Each participant will walk at 70 % of his/her VO2max for 20 minutes on treadmill.
Drug: Metoprolol Succinate ER — Each participant will receive metoprolol succinate starting at 50mg/day, titrated bi-weekly up to 200 mg/day for total duration of 6 weeks.

SUMMARY:
The purpose of the study is to understand the origins of differential response to beta-blockers in African-Americans and may provide insight regarding racial differences in cardiovascular risk.

DETAILED DESCRIPTION:
The heart is an endocrine organ. The natriuretic peptides are hormones produced in the heart and are secreted in response to increased wall stress in atria and ventricles. The principal circulating NPs are Atrial Natriuretic Peptide (ANP) and B-type Natriuretic Peptide (BNP). The endocrine actions of NPs are natriuresis and dilatation of peripheral arteries.

The NPs concentrations are elevated in heart failure (HF) and hypertension (HTN) due to volume and pressure overload. Therefore, NPs are used as diagnostic and prognostic markers in heart failure. However, NPs role in healthy individuals is not known.

Previous studies have shown that reduced NP levels are associated with a greater risk of HTN. Moreover, African-Americans have lower resting NP levels than Caucasians. We hypothesize that relative NP deficiency in African American compared to Caucasian has the potential to contribute to increase risk of all-cause mortality, HTN, HF and its sequelae.

Evidence from multiple clinical trials has positioned beta-blockers as a standard heart failure therapy. Beta-blocker therapy leads to increased NP levels and suppression of Renin-aldosterone-angiotensin system (RAAS) system. Suppression of renin levels by beta-blockers has been shown as a potential mechanism of benefit in HF. However, study shows that beta-blockers are less effective in African-Americans compared to Caucasians in HF treatment. So, the investigators have proposed a pilot study to look for race-based differences in the NP and RAAS response to metoprolol in healthy individuals.

Additionally, exercise has been reported to increase NP levels. ANP increases more than BNP with exercise. But there is no data of NP changes in African-American with exercise. So the investigators have proposed a sub-study of race-based difference in ANP and BNP response to exercise.

40 African-American and 40 Caucasians normotensive or pre-hypertensive (healthy) individuals will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 40 years
* Blood pressure less than 140/90 mm Hg
* Able to perform exercise capacity test
* BMI 18-30 kg/m2
* Willing to adhere to study drug

Exclusion Criteria:

* History of cardiovascular disease or use of medications for CVD
* History of hypertension or use of BP lowering medications
* Blood pressure less than 100/60 mm Hg
* Heart rate less than 60 beats/min
* Depression
* Diabetes or use of anti-diabetic medications
* Renal disease (eGFR < 60ml/min/1.73m2)
* Current or prior smokers
* Pregnant or use of Hormone Replacement Therapy (HRT) or oral contraceptives (OCP) or steroids

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2017-04-30 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pankaj Arora, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Davis ME, Richards AM, Nicholls MG, Yandle TG, Frampton CM, Troughton RW. Introduction of metoprolol increases plasma B-type cardiac natriuretic peptides in mild, stable heart failure. Circulation. 2006 Feb 21;113(7):977-85. doi: 10.1161/CIRCULATIONAHA.105.567727. Epub 2006 Feb 13. PMID 16476851
- [Result] Trowbridge CA, Gower BA, Nagy TR, Hunter GR, Treuth MS, Goran MI. Maximal aerobic capacity in African-American and Caucasian prepubertal children. Am J Physiol. 1997 Oct;273(4):E809-14. doi: 10.1152/ajpendo.1997.273.4.E809. PMID 9357812
- [Result] Hunter GR, Weinsier RL, McCarthy JP, Enette Larson-Meyer D, Newcomer BR. Hemoglobin, muscle oxidative capacity, and VO2max in African-American and Caucasian women. Med Sci Sports Exerc. 2001 Oct;33(10):1739-43. doi: 10.1097/00005768-200110000-00019. PMID 11581560
- [Result] Steele IC, McDowell G, Moore A, Campbell NP, Shaw C, Buchanan KD, Nicholls DP. Responses of atrial natriuretic peptide and brain natriuretic peptide to exercise in patients with chronic heart failure and normal control subjects. Eur J Clin Invest. 1997 Apr;27(4):270-6. doi: 10.1046/j.1365-2362.1997.1070653.x. PMID 9134374
- [Result] Shetty NS, Gaonkar M, Patel N, Vekariya N, Yerabolu K, Dhaliwal JS, Buford TW, Gower B, Li P, Wang TJ, Arora G, Arora P. Differences in natriuretic peptide response in self-identified white and black individuals: a physiological clinical trial. Nat Commun. 2025 Feb 13;16(1):1621. doi: 10.1038/s41467-024-55648-2. PMID 39948072

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Black Participants | White Participants
Started | 40 | 40
Completed | 40 | 40
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Black Participants | White Participants | Total
Number analyzed (Participants) | 40 | 40 | 80
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 27 [22 to 32] | 25 [20 to 30] | 26 [21 to 30]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 19 | 40
  Male | 19 | 21 | 40
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 40 | 40 | 80
  Unknown or Not Reported | 0 | 0 | 0
Body Mass Index (BMI) [Median (Inter-Quartile Range); unit: kg/m²] | 25.1 [22.4 to 27.7] | 24.1 [22.4 to 26.8] | 24.5 [22.4 to 27.6]
Systolic Blood Pressure (SBP) [Median (Inter-Quartile Range); unit: mmHg] | 109 [105 to 116] | 108 [102 to 116] | 109 [103 to 117]
Diastolic Blood Pressure (DBP) [Median (Inter-Quartile Range); unit: mmHg] | 67 [64 to 74] | 70 [63 to 75] | 69 [63 to 75]
Heart Rate [Median (Inter-Quartile Range); unit: beats per minute] | 69 [63 to 77] | 70 [62.7 to 79] | 70 [63 to 78]
Fasting Glucose [Median (Inter-Quartile Range); unit: mg/dL] | 83.0 [80.0 to 89.0] | 86.5 [79.0 to 90.0] | 85.0 [80.0 to 90.0]
Hemoglobin [Median (Inter-Quartile Range); unit: g/dL] | 13.3 [12.5 to 14.1] | 14.1 [12.6 to 14.8] | 13.5 [12.6 to 14.6]
Insulin [Median (Inter-Quartile Range); unit: mg/dL] | 6.5 [3.9 to 9.0] | 5.9 [3.7 to 7.9] | 6.2 [3.9 to 8.5]
Creatinine [Median (Inter-Quartile Range); unit: mg/dL] | 1.0 [0.8 to 1.1] | 0.9 [0.7 to 1.0] | 0.9 [0.7 to 1.0]
Aspartate Aminotransferase (AST) [Median (Inter-Quartile Range); unit: U/L] | 17.0 [15.0 to 25.0] | 17.0 [14.5 to 21.0] | 17.0 [15.0 to 22.0]
Alanine Aminotransferase (ALT) [Median (Inter-Quartile Range); unit: U/L] | 14.0 [11.0 to 18.0] | 14.5 [12.0 to 20.5] | 14.0 [12.0 to 20.0]
Midregional pro- Atrial Natriuretic Peptide (MRproANP) [Median (Inter-Quartile Range); unit: pmol/L] | 43 [31 to 56] | 47 [35 to 58] | 44 [32 to 57]
B-type Natriuretic Peptide (BNP) [Median (Inter-Quartile Range); unit: ng/L] | 16.0 [11.0 to 25.0] | 15.0 [9.0 to 27.0] | 15.0 [10.0 to 25.0]
N-terminal pro-Btype Natriuretic Peptide (NTproBNP) [Median (Inter-Quartile Range); unit: ng/L] | 17 [6 to 31] | 20 [13 to 39] | 19 [9 to 34]
Left Ventricular Hypertrophy [Number; unit: Percentage of Participants] — Left Ventricular Hypertrophy (LVH) was assessed using the Minnesota coding criteria for high amplitude R waves. Criteria include: (1) R amplitude > 26 mm in leads V5 or V6, or > 20 mm in leads I, II, III, aVF; or R amplitude > 12 mm in lead aVL; (2) Right R amplitude ≥ 5 mm and R ≥ S amplitude in the majority of beats in lead V1, with R amplitude located to the left of V1; or (3) R amplitude > 15 mm but ≤ 20 mm in lead I, or R amplitude in leads V5 or V6 plus S amplitude in lead V1 > 35 mm. All amplitudes were measured from the second-to-last complete normal beat. Population: Cardiac function parameters where only collected for a limited number of participants
  Percentage of Participants
    number analyzed (Participants) | 21 | 30 | 51
    (all) | 0.0 | 6.7 | 3.9
Left Atrial Enlargement [Number; unit: Percentage of Participants] — Left Atrial Enlargement (LAE) was assessed using electrocardiographic (ECG) criteria. Criteria include: (1) In lead II: presence of a bifid P wave with > 40 ms between the two peaks or a total P wave duration > 110 ms; (2) In lead V1: presence of a biphasic P wave with a terminal negative portion lasting > 40 ms, or a terminal negative portion > 1 mm in depth. These criteria were used to identify LAE based on ECG analysis. Population: Cardiac function parameters where only collected for a limited number of participants
  Percentage of Participants
    number analyzed (Participants) | 21 | 30 | 51
    (all) | 4.8 | 23.3 | 15.7

OUTCOME MEASURES:

1. Primary Outcome: Change in Plasma BNP After 6-weeks of Beta-Blocker
Description: Mean percentage change in plasma BNP concentrations in response to 6 weeks of Beta-Blocker between Black participants and White participants
Time Frame: 6 weeks
Measure: Mean (95% Confidence Interval); unit: Percentage Change in Plasma BNP levels
Arm/Group | Black Participants | White Participants
Number analyzed (Participants) | 40 | 40
Percentage Change in Plasma BNP levels | 45 [7 to 95] | 74 [30 to 133]

2. Primary Outcome: Change in Plasma NT-proBNP After 6-weeks of Beta-Blocker
Description: Mean percentage change in plasma NT-proBNP concentrations in response to 6 weeks of Beta-Blocker between Black participants and White participants
Time Frame: 6 weeks
Measure: Mean (95% Confidence Interval); unit: Percentage Change in Plasma NT-proBNP
Arm/Group | Black Participants | White Participants
Number analyzed (Participants) | 40 | 40
Percentage Change in Plasma NT-proBNP | 95 [31 to 190] | 99 [35 to 193]

3. Primary Outcome: Change in Plasma MR-proANP After 6-weeks of Beta-Blocker
Description: Mean percentage change in plasma MR-proANP concentrations in response to 6 weeks of Beta-Blocker between Black participants and White participants
Time Frame: 6 weeks
Measure: Mean (95% Confidence Interval); unit: Percentage Change in Plasma MR-proANP
Arm/Group | Black Participants | White Participants
Number analyzed (Participants) | 40 | 40
Percentage Change in Plasma MR-proANP | 18 [-5 to 47] | 16 [-6 to 44]

4. Secondary Outcome: Change in Plasma BNP After Standardized Exercise Challenge
Description: Mean percentage change in plasma BNP concentrations in response to exercise
Time Frame: Mean percentage change in plasma BNP concentrations from baseline to 20 minutes post-exercise (immediately after exercise)
Measure: Mean (95% Confidence Interval); unit: Percentage change in Plasma BNP
Arm/Group | Black Participants | White Participants
Number analyzed (Participants) | 40 | 40
Percentage change in Plasma BNP | 59 [14 to 114] | 61 [20 to 116]

5. Secondary Outcome: Change in Plasma NT-proBNP After Standardized Exercise Challenge
Description: Mean percentage change in plasma NT-proBNP concentrations in response to exercise
Time Frame: Mean percentage change in plasma NT-proBNP concentrations from baseline to 20 minutes post-exercise (immediately after exercise)
Measure: Mean (95% Confidence Interval); unit: Percentage change in Plasma NT-proBNP
Arm/Group | Black Participants | White Participants
Number analyzed (Participants) | 40 | 40
Percentage change in Plasma NT-proBNP | 11 [-28 to 69] | 23 [20 to 87]

6. Secondary Outcome: Change in Plasma MR-proANP After Standardized Exercise Challenge
Description: Mean percentage change in plasma MR-proANP concentrations in response to exercise
Time Frame: Mean percentage change in plasma MR-proANP concentrations from baseline to 20 minutes post-exercise (immediately after exercise)
Measure: Mean (95% Confidence Interval); unit: Percentage change in Plasma MR-proANP
Arm/Group | Black Participants | White Participants
Number analyzed (Participants) | 40 | 40
Percentage change in Plasma MR-proANP | 35 [8 to 68] | 43 [15 to 78]

ADVERSE EVENTS:
Time Frame: Adverse events were collected after the completion of the screening visit, during the exercise visits, and during the Beta-Blocker intervention period for a total of 14 weeks
Arm/Group | Black Participants | White Participants
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 6/40 | 7/40
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Black Participants (N=40) | White Participants (N=40)
Headache (Nervous system disorders) | 6 (6) | 7 (7)
Nausea (Gastrointestinal disorders) | 5 (5) | 6 (6)
Vasovagal Response (Nervous system disorders) | 2 (2) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-01-18): https://cdn.clinicaltrials.gov/large-docs/84/NCT03070184/Prot_SAP_005.pdf
  • Informed Consent Form (2023-01-18): https://cdn.clinicaltrials.gov/large-docs/84/NCT03070184/ICF_002.pdf